CLINICAL TRIAL: NCT04907513
Title: Amotivational Syndrome and Fatigue in Neurosurgery: The Impact of Neuroinflammation
Brief Title: Amotivational Syndrome and Fatigue in Neurosurgery
Acronym: DENI-CARE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: PBN_2021_1
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Cerebral Injury; Motivation; Fatigue
Keywords: cerebrospinal fluid
MeSH Terms: conditions — Brain Injuries; Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Amotivational Syndrome: Patients required an external drainage of the cerebrospinal fluid.
  Interventions: Other: Assessment of the Motivational State

INTERVENTIONS:
Other: Assessment of the Motivational State — A motivational interviewing algorithm developed in Rothschild Hospital for this study will be used. The results range between 0% (worst motivational state) to 100% (best motivational state).

SUMMARY:
Depression is a major public concern associated with profound distress, intense suffering, and impairment in social, professional and familial functioning. Among the numerous symptoms defining depression, fatigue and motivation are not only frequent but also highly associated with poor quality of life and resistance to conventional antidepressant. Recent data, mainly obtained in animals, suggest that these symptoms may be linked to inflammatory processes within the central nervous system. Yet access to the brain is too invasive for exploring this link in patients with psychiatric conditions. However, certain conditions in neurosurgery, such as aneurysm rupture, require external evacuation, over several days or weeks, of the fluid bathing the brain through a catheter directly inserted into it. Critically, these patients also exhibit extreme exhaustion and fluctuating motivation, allowing to investigate the involvement of neuroinflammation in lack of motivation and fatigue by carrying out repeated motivation assessments with short behavioral tests (around ten minutes), while performing an analysis of inflammation markers in the fluid evacuated from the brain. The identification of inflammatory mechanisms underlying lack of motivation and fatigue could lead to the development of treatments for both resistant depression and motivation deficits that largely hamper rehabilitation in neurosurgery.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years old
* Patients required an external cerebrospinal fluid drainage

Exclusion Criteria:

* Pregnant or breast feeding patient
* Patient under legal protection
* Patient opposition to participate in this study

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients required an external drainage of the cerebrospinal fluid
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2021-12-04 (Actual); Primary Completion 2023-12-04 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Nerotransmitter levels in cerebrospinal fuid in relation to patient motivational condition | 36 months
  Study the correlation between serotonin, dopamin and glutamate concentrations in the cerebrospinal fluid with the motivational state of the patients

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Fondation Adolphe de Rothschild, Paris, Île-de-France Region, France